CLINICAL TRIAL: NCT02406183
Title: Phase I Trial of Stereotactic Body Radiotherapy With Concurrent Fixed Dose Immune Checkpoint Inhibitors in Metastatic Melanoma: Dose Limiting Toxicity and Abscopal Effect
Brief Title: Trial of SBRT With Concurrent Ipilimumab in Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radiotherapie (Other)
Responsible Party: Sponsor-Investigator, Radiotherapie, MD, PhD, University Hospital, Ghent
Organization: University Hospital, Ghent (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC 2015/0025
Record Dates: First submitted 2015-03-17; First posted 2015-04-02 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Melanoma; Effects of Immunotherapy; Adverse Effect of Radiation Therapy
MeSH Terms: conditions — Melanoma; Radiation Injuries | interventions — Radiosurgery; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (SBRT, Ipilimumab) (Experimental): Drug: Ipilimumab Dosage: Ipilimumab will be administered intravenously at 3 mg/kg every 3 weeks for 4 cycles,
  Radiation: Stereotactic Body Radiotherapy Radiation therapy 24 Grays in 8 Grays fractions, Radiation therapy 30 Grays in 10 Grays fractions, Radiation therapy 36 Grays in 12 Grays fractions
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT); Drug: Ipilimumab

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy (SBRT) — The SBRT dose will be escalated in 3 steps as described above and will be given on d39, d41 and d43
  Other Names: SABR
Drug: Ipilimumab — Ipilimumab 3mg/kg will be given IV on d1, d22, d43 and d64
  Other Names: Yervoy

SUMMARY:
The prognosis of advanced metastatic melanoma remains poor although a breakthrough has been achieved with the novel anti-CTLA-4 treatment (ipilimumab) for a subset of patients. Unfortunately, due to immune resistance, the majority of patients do not obtain long-lasting clinical benefit. Radiotherapy is able to interfere with immune resistance by inducing immunogenic cell death. Preclinical evidence indicates that combining radiotherapy with anti-CTLA-4 treatment increases response rates compared to single agent treatment. These data are supported by several spectacular clinical cases and one retrospective study. The investigators hypothesize that combining ipilimumab with radiotherapy will result in a higher response rate compared to ipilimumab or radiotherapy in monotherapy. Given the complexity of the interaction in anti-tumor immunity, the first goal of this project is to assess the safety of the combined treatment.

DETAILED DESCRIPTION:
The safety profiles of ipilimumab and SBRT are well studied separately 22-24, but prospective data on the combination of ipilimumab and high-dose SBRT are lacking. Consequently, the first goal of the proposed prospective phase I trial is to assess the safety (dose limiting toxicity, DLT) of the combination of high-dose SBRT and ipilimumab in patients with advanced melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and willingness to comply to the treatment and follow-up
* Histological diagnosis of melanoma,
* at least 3 extracranial measurable metastatic lesions per RECIST 1.1,
* Karnofsky Performance score >60,
* Age ≥18,
* Life expectancy ≥ 16 weeks
* Women of childbearing potential must have a negative serum pregnancy test within 14 days of first dose of study treatment. Men and women should agree to use effective contraception, during the study and for 1 month following the last dose of investigational product.
* ≥ 28 days between last treatment with standard or experimental chemotherapy, surgery, radiotherapy, cytokine therapy or immunotherapy. Patient should be completely recuperated of any clinical toxicity developed during previous treatments.
* Patients should have adequate organ function for ipilimumab treatment

Exclusion Criteria:

* Central nervous system (CNS) metastases at baseline, with the exception of those subjects who have previously-treated CNS metastases (surgery ± radiotherapy, radiosurgery, or gamma knife) and who meet both of the following criteria: a) are asymptomatic and b) have no requirement for steroids or enzyme-inducing anticonvulsants.
* Prior malignancy: Subjects who have had another malignancy and have been disease-free for 5 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible
* Prior radiotherapy preventing treatment with SBRT.
* Disorder precluding understanding of trial information.
* Autoimmune disease: Patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) and autoimmune disorders such as rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus or autoimmune vasculitis [e.g., Wegener's Granulomatosis] are excluded from this study.
* Known Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C.
* Concomitant therapy with any of the following: IL-2, interferon or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigational therapies; or chronic use of systemic corticosteroids (used in the management of cancer or non-cancer-related illnesses).
* Pregnant women
* Breast feeding
* History of or current immunodeficiency disease or prior treatment compromising immune function, prior allogeneic stem cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Maximal tolerated dose (MDT) that is associated with dose-limiting toxicity (DLT) in 25% of patients. | 2 years

SECONDARY OUTCOMES:
Preliminary anti-tumor activity following escalating doses of radiation combined to ipilimumab using the immune related response criteria irRC | 2 years
Overall survival | 2 years
Progression-free survival | 2 years
Immunomonitoring (absolute lymphocyte count) | 2 years
  absolute lymphocyte count
Immunomonitoring (frequencies of Foxp3+ Treg-cells) | 2 years
  frequencies of Foxp3+ Treg-cells
Immunomonitoring (functional analysis looking at shifts in Th1/Th2/Th17) | 2 years
  functional analysis looking at shifts in Th1/Th2/Th17
Immunomonitoring (plasmacytoid dendritic cells and myeloid derived suppressor cells and their IDO expression) | 2 years
  plasmacytoid dendritic cells and myeloid derived suppressor cells and their IDO expression,

CONTACTS AND LOCATIONS:
Overall Officials: Piet Ost, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Dept. of Radiotherapy, Ghent University Hospital, Ghent, Oost-Vlaanderen, Belgium